CLINICAL TRIAL: NCT02526732
Title: Influence of Hepatic Inflammation and Hepatocellular Apoptosis on Physical Performance and Training Effect in Patients With Non - Alcoholic Steatohepatitis
Brief Title: Hepatic Inflammation and Physical Performance in Patients With NASH
Acronym: HELP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Priv.-Doz. Dr. J. Schattenberg (Other)
Responsible Party: Sponsor-Investigator, Priv.-Doz. Dr. J. Schattenberg, Prov.-Doz. Dr. med., Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015_04_001_HELP
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: NASH; fatty Liver; VO2 max; M30 antigen
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- individual training program (Experimental): Patients will be offered an individual training program. Physical performance and surrogate parameters of liver inflammation will assessed in physical examinations before and after the training phase.
  Interventions: Other: individual training program

INTERVENTIONS:
Other: individual training program — Training period of 8 weeks: Independently running exercises for 30-45 minutes two to three times a week. Every two weeks group training sessions are offered accompanied by a sports physician.

SUMMARY:
The aim of the study is to examine the influence of hepatic inflammation or damage on physical performance (maximal oxygen uptake, VO2max) depending on the histologic state of the liver. The study population are patients with fatty liver disease and non-alcoholic steatohepatitis (NASH). All study participants obtain an individual training plan with individual and group training sessions for a period of 8 weeks. At the beginning and end of the training phase a sport physiological examination is carried out. In the study group the effect of regular examinations is surveyed by surrogate parameters of liver inflammation.

DETAILED DESCRIPTION:
The study is planned over a period of 24 months. Study participants should be twice examined sport physiologically in a period of 12 weeks. In the study group the influence of regular exercise on surrogate parameters of liver inflammation is investigated over a study period of 8 weeks. Before the exercise all study participants are subjected to a first physiological examination (about 3 hours). This includes a physical examination with detection of body weight, waist circumference and body fat analysis, venous blood, oral glucose tolerance test, ultrasonography of the liver and determination of endothelial function (flow-mediated vasodilatation, FMD) by Doppler analysis. Within 4 weeks after the first examination a sport physical examination is carried out at the Institute of Sports Science at the University of Mainz. This examination contains identification of physical fitness and individual lactate performance diagnostics. In addition, indirect calorimetry is carried out under exercise conditions using spiroergometry to determine the maximal oxygen uptake (VO2max) with special emphasis on the fat metabolism rate at low physical activity. Subsequently to the examination an 8-week training period based on individual training / performance plans is followed. The training plans include independently running exercises for 30-45 minutes two to three times a week. Every two weeks group training sessions are offered accompanied by a sports physician. Within the planed four groups training sessions blood samples will be taken to determinate free circulating DNA and assess lactate values under exercise conditions. After the training phase, a second sport physical examination including physical performance and a final physiological examination including surrogate parameters of liver inflammation are carried out. For statistical analysis, the physical performance of the study participants is examined. Hence patients with histologically proven NASH (NAS score) and confirmed inflammation (increased M30 antigen) are compared to age and gender matched patients with histologically proven fatty liver without inflammation reaction as well as to retrospective data of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven NASH or fatty liver disease

Exclusion Criteria:

* bariatric surgery within the last 5 years
* BMI< 18,5 kg/m2 or > 45 kg/m2
* heart attack or stroke within the last 6 months
* higher-grade coronary artery disease (CAD III-IV)
* chronic obstructive pulmonary disease (asthma , COPD)
* renal insufficiency
* uncontrolled hypertension or metabolic abnormalities
* alcohol consumption > 30 g / day (male) and > 20 g / day (female)
* pregnancy
* concomitant medication able to cause a secondary NASH (eg tamoxifen , corticosteroids )
* concomitant medication able to affect inflammation (eg TNF antagonists)
* concomitant anticoagulant medication (eg phenprocoumon, NOAC)
* other immunological or inflammatory diseases (eg, systemic lupus erythematosus)
* musculoskeletal disorders, preventing sport physiological investigations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Change in physical performance | 0-8 weeks
  Change of Vo2max from week 0 to week 8

SECONDARY OUTCOMES:
Change in liver inflammation | 8 weeks
  Change of NAS score at week 0 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Galle, MD, Study Director — I. Medizinische Klinik und Poliklinik, Universitätsmedizin Mainz
Locations (1):
- University Medical Center of the Johannes Gutenber Univeristy, Mainz, Germany

IPD SHARING:
Plan to Share IPD: Yes
Publication in scientific journals and conferences

REFERENCES:
- [Background] Clark JM. The epidemiology of nonalcoholic fatty liver disease in adults. J Clin Gastroenterol. 2006 Mar;40 Suppl 1:S5-10. doi: 10.1097/01.mcg.0000168638.84840.ff. PMID 16540768
- [Background] Blachier M, Leleu H, Peck-Radosavljevic M, Valla DC, Roudot-Thoraval F. The burden of liver disease in Europe: a review of available epidemiological data. J Hepatol. 2013 Mar;58(3):593-608. doi: 10.1016/j.jhep.2012.12.005. PMID 23419824
- [Background] Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther. 2011 Aug;34(3):274-85. doi: 10.1111/j.1365-2036.2011.04724.x. Epub 2011 May 30. PMID 21623852
- [Background] Sanyal AJ. NASH: A global health problem. Hepatol Res. 2011 Jul;41(7):670-4. doi: 10.1111/j.1872-034X.2011.00824.x. PMID 21711426
- [Background] Mehal WZ. The Gordian Knot of dysbiosis, obesity and NAFLD. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):637-44. doi: 10.1038/nrgastro.2013.146. Epub 2013 Aug 20. PMID 23958600
- [Background] Schattenberg JM, Schuppan D. Nonalcoholic steatohepatitis: the therapeutic challenge of a global epidemic. Curr Opin Lipidol. 2011 Dec;22(6):479-88. doi: 10.1097/MOL.0b013e32834c7cfc. PMID 22002020
- [Background] Fargion S, Porzio M, Fracanzani AL. Nonalcoholic fatty liver disease and vascular disease: state-of-the-art. World J Gastroenterol. 2014 Oct 7;20(37):13306-24. doi: 10.3748/wjg.v20.i37.13306. PMID 25309067
- [Background] Krasnoff JB, Painter PL, Wallace JP, Bass NM, Merriman RB. Health-related fitness and physical activity in patients with nonalcoholic fatty liver disease. Hepatology. 2008 Apr;47(4):1158-66. doi: 10.1002/hep.22137. PMID 18266250
- [Background] Noakes TD. Maximal oxygen uptake: "classical" versus "contemporary" viewpoints: a rebuttal. Med Sci Sports Exerc. 1998 Sep;30(9):1381-98. doi: 10.1097/00005768-199809000-00007. PMID 9741607
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Background] Sreenivasa Baba C, Alexander G, Kalyani B, Pandey R, Rastogi S, Pandey A, Choudhuri G. Effect of exercise and dietary modification on serum aminotransferase levels in patients with nonalcoholic steatohepatitis. J Gastroenterol Hepatol. 2006 Jan;21(1 Pt 1):191-8. doi: 10.1111/j.1440-1746.2005.04233.x. PMID 16706832
- [Background] Fealy CE, Haus JM, Solomon TP, Pagadala M, Flask CA, McCullough AJ, Kirwan JP. Short-term exercise reduces markers of hepatocyte apoptosis in nonalcoholic fatty liver disease. J Appl Physiol (1985). 2012 Jul;113(1):1-6. doi: 10.1152/japplphysiol.00127.2012. Epub 2012 May 10. PMID 22582214
- [Background] Bae JC, Suh S, Park SE, Rhee EJ, Park CY, Oh KW, Park SW, Kim SW, Hur KY, Kim JH, Lee MS, Lee MK, Kim KW, Lee WY. Regular exercise is associated with a reduction in the risk of NAFLD and decreased liver enzymes in individuals with NAFLD independent of obesity in Korean adults. PLoS One. 2012;7(10):e46819. doi: 10.1371/journal.pone.0046819. Epub 2012 Oct 22. PMID 23110056
- [Background] Kistler KD, Brunt EM, Clark JM, Diehl AM, Sallis JF, Schwimmer JB; NASH CRN Research Group. Physical activity recommendations, exercise intensity, and histological severity of nonalcoholic fatty liver disease. Am J Gastroenterol. 2011 Mar;106(3):460-8; quiz 469. doi: 10.1038/ajg.2010.488. Epub 2011 Jan 4. PMID 21206486
- [Background] Swain MG. Fatigue in liver disease: pathophysiology and clinical management. Can J Gastroenterol. 2006 Mar;20(3):181-8. doi: 10.1155/2006/624832. PMID 16550262
- [Background] Brun P, Castagliuolo I, Di Leo V, Buda A, Pinzani M, Palu G, Martines D. Increased intestinal permeability in obese mice: new evidence in the pathogenesis of nonalcoholic steatohepatitis. Am J Physiol Gastrointest Liver Physiol. 2007 Feb;292(2):G518-25. doi: 10.1152/ajpgi.00024.2006. Epub 2006 Oct 5. PMID 17023554
- [Background] Wigg AJ, Roberts-Thomson IC, Dymock RB, McCarthy PJ, Grose RH, Cummins AG. The role of small intestinal bacterial overgrowth, intestinal permeability, endotoxaemia, and tumour necrosis factor alpha in the pathogenesis of non-alcoholic steatohepatitis. Gut. 2001 Feb;48(2):206-11. doi: 10.1136/gut.48.2.206. PMID 11156641
- [Background] Miura K, Ohnishi H. Role of gut microbiota and Toll-like receptors in nonalcoholic fatty liver disease. World J Gastroenterol. 2014 Jun 21;20(23):7381-91. doi: 10.3748/wjg.v20.i23.7381. PMID 24966608
- [Background] Zhu L, Baker SS, Gill C, Liu W, Alkhouri R, Baker RD, Gill SR. Characterization of gut microbiomes in nonalcoholic steatohepatitis (NASH) patients: a connection between endogenous alcohol and NASH. Hepatology. 2013 Feb;57(2):601-9. doi: 10.1002/hep.26093. Epub 2013 Jan 8. PMID 23055155
- [Derived] Huber Y, Pfirrmann D, Gebhardt I, Labenz C, Gehrke N, Straub BK, Ruckes C, Bantel H, Belda E, Clement K, Leeming DJ, Karsdal MA, Galle PR, Simon P, Schattenberg JM. Improvement of non-invasive markers of NAFLD from an individualised, web-based exercise program. Aliment Pharmacol Ther. 2019 Oct;50(8):930-939. doi: 10.1111/apt.15427. Epub 2019 Jul 25. PMID 31342533
- [Derived] Pfirrmann D, Huber Y, Schattenberg JM, Simon P. Web-Based Exercise as an Effective Complementary Treatment for Patients With Nonalcoholic Fatty Liver Disease: Intervention Study. J Med Internet Res. 2019 Jan 2;21(1):e11250. doi: 10.2196/11250. PMID 30602434
- [Derived] Pfirrmann D, Haller N, Huber Y, Jung P, Lieb K, Gockel I, Poplawska K, Schattenberg JM, Simon P. Applicability of a Web-Based, Individualized Exercise Intervention in Patients With Liver Disease, Cystic Fibrosis, Esophageal Cancer, and Psychiatric Disorders: Process Evaluation of 4 Ongoing Clinical Trials. JMIR Res Protoc. 2018 May 22;7(5):e106. doi: 10.2196/resprot.8607. PMID 29789277